CLINICAL TRIAL: NCT00512252
Title: A Phase I/II Study of AMD3100 With Mitoxantrone, Etoposide and Cytarabine (AMD3100+MEC) in Relapsed or Refractory AML
Brief Title: AMD3100 Plus Mitoxantrone, Etoposide and Cytarabine in Acute Myeloid Leukemia
Acronym: AMD3100+MEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0227 / 201011796
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Plerixafor; CXCR4; Chemosensitization
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — plerixafor; Mitoxantrone; Etoposide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I Dose Escalation (Experimental): * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 1 AMD3100 dose = 80 mcg/kg/d
  Dose Level 2 AMD3100 dose = 160 mcg/kg/d
  Interventions: Drug: AMD3100; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Phase II Dose Treatment (Experimental): * AMD 3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 3 AMD3100 dose=240 mcg/kg/d (this was the Phase II dose)
  Interventions: Drug: AMD3100; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: AMD3100
  Other Names: Plerixafor
Drug: Mitoxantrone
  Other Names: Novantrone
Drug: Etoposide
  Other Names: VP-16; Vepesid; Etopophos
Drug: Cytarabine
  Other Names: Ara-C; Cytosar-U; Tarabine PFS

SUMMARY:
This study is a phase I/II study to determine the safety and efficacy of AMD3100 when combined with mitoxantrone, etoposide, and cytarabine in patients with relapsed or refractory AML.

We hypothesize that disrupting the interaction between AML blasts and the marrow microenvironment with AMD3100 may enhance the cytotoxic effect of chemotherapy.

DETAILED DESCRIPTION:
The interaction of leukemic blasts with the bone marrow microenvironment is postulated to be an important mediator of chemoresistance in AML. Although a number of receptor / ligand pairs have been implicated, the CXCR4 / SDF-1 axis functions as the principal regulator of homing and retention of both normal and malignant hematopoietic cells in the marrow. AMD3100 is a bicyclam molecule which reversibly blocks CXCR4 binding to SDF-1 and is being developed clinically as a mobilization agent for hematopoietic stem cell transplantation. Preclinical data from our group has demonstrated that in murine models, plerixafor can disrupt the interaction of leukemic cells with the marrow microenvironment and sensitize blasts to the effect of chemotherapy. Based on these data, we have initiated a phase I/II study in patients with relapsed or refractory AML in which plerixafor is administered prior to salvage chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia diagnosed by WHO criteria with one of the following:

   1. Primary refractory disease following >= 1 rounds of induction chemotherapy
   2. First relapse or higher
2. Age between 18 and 70 years of age
3. Adequate organ function defined as Creatinine <= 1.5 x institutional ULN; AST, ALT, total bilirubin <= 2 x ULN; Left ventricular ejection fraction of >= 40% by MUGA scan
4. Women of childbearing potential and sexually active males must be willing and able to use effective contraception while on study
5. Able to provide signed informed consent prior to registration on study

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML with t(15;17)(q22;q11) and variants)
2. Peripheral blood blast count > 20 x 103 /mm3
3. Active CNS involvement with leukemia
4. Previous treatment with MEC or other regimen containing both mitoxantrone and etoposide
5. Pregnant or nursing
6. Receiving any other investigational agent
7. Colony stimulating factors filgrastim, pegfilgrastim or sargramostim within 2 weeks of study
8. Less than 2 weeks from the completion of any previous cytotoxic chemotherapy
9. Severe concurrent illness that would limit compliance with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L. Uy, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Uy GL, Rettig MP, Motabi IH, McFarland K, Trinkaus KM, Hladnik LM, Kulkarni S, Abboud CN, Cashen AF, Stockerl-Goldstein KE, Vij R, Westervelt P, DiPersio JF. A phase 1/2 study of chemosensitization with the CXCR4 antagonist plerixafor in relapsed or refractory acute myeloid leukemia. Blood. 2012 Apr 26;119(17):3917-24. doi: 10.1182/blood-2011-10-383406. Epub 2012 Feb 2. PMID 22308295
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 07/12/2007 until 01/14/2010.
Groups:
- Phase I Dose Escalation (Dose Level 1): * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 1 AMD3100 dose = 80 mcg/kg/d
- Phase I Dose Escalation (Dose Level 2): * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 2 AMD3100 dose = 160 mcg/kg/d
- Phase II Dose Treatment (Dose Level 3): * AMD 3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 3 AMD3100 dose=240 mcg/kg/d (this was the Phase II dose).
  The 6 participants that were enrolled in Dose Level 3 in the Phase I portion of the study were carried over to the Phase II analysis. 40 additional patients were enrolled in the Phase II portion of the study using the Dose Level 3 dose.
Period: Overall Study
Arm/Group | Phase I Dose Escalation (Dose Level 1) | Phase I Dose Escalation (Dose Level 2) | Phase II Dose Treatment (Dose Level 3)
Started | 3 | 3 | 46
Completed | 3 | 3 | 43
Not Completed | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The 6 participants that were enrolled in Dose Level 3 in the Phase I portion of the study were carried over to the Phase II analysis. 40 additional patients were enrolled in the Phase II portion of the study using the Dose Level 3 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation (Dose Level 1) | Phase I Dose Escalation (Dose Level 2) | Phase II Dose Treatment (Dose Level 3) | Total
Number analyzed (Participants) | 3 | 3 | 46 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 3 | 3 | 40 | 46
  >=65 years | 0 | 0 | 5 | 5
Age, Continuous [Median (Full Range); unit: years] | 58 [44 to 62] | 24 [22 to 39] | 51 [18 to 71] | 51 [18 to 71]
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 26 | 30
  Male | 1 | 1 | 20 | 22
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 46 | 52
Acute myeloid leukemia (AML) source [Number; unit: participants] — MDS = myelodysplastic syndrome MPD = myeloproliferative disease
  participants
    De novo AML | 3 | 2 | 36 | 41
    Therapy related | 0 | 1 | 4 | 5
    Prior MDS/MPD | 0 | 0 | 6 | 6
Prior transplantation [Number; unit: participants]
  Autologous | 0 | 0 | 3 | 3
  Allogeneic | 0 | 0 | 6 | 6
  No prior transplant | 3 | 3 | 37 | 43
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Grade 0 Fully active able to carry on all predisease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (light house work/office work)
  2. Ambulatory, capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours
  3. Capable of limited selfcare, confined to bed/chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on selfcare. Totally confined to bed/chair
  5. Dead
  participants
    0 | 2 | 2 | 25 | 29
    1 | 1 | 1 | 10 | 12
    2 | 0 | 0 | 3 | 3
    Unknown | 0 | 0 | 8 | 8
Treatment Indication [Number; unit: participants]
  First relapse, first salvage | 3 | 2 | 32 | 37
  Primary refractory | 0 | 1 | 10 | 11
  >=Second relapse/salvage | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only: Optimal Dose of AMD3100 Plus MEC in Patients With Relapsed or Refractory AML
Description: A standard 3+3 design was used in the Phase I portion starting with the AMD3100 dose of 80 mcg/kg and escalating by 80 mcg/kg for each successive cohort up to a maximum of 240 mcg/kg/d. The optimal dose was defined as the highest dose of AMD3100 <= 240 mcg/kg at which 0-1 of 6 patients experienced a dose limiting toxicity.
Time Frame: Completion of all patients in Phase I portion (232 days)
Population: The Phase I Dose Escalation portion included (3) patients enrolled in Dose Level 1 and (3) patients enrolled in Dose Level 2. The (6) patients enrolled in Dose Level 3 that determined the Phase II dose are included in the population for this outcome.
Measure: Number; unit: mcg/kg
Groups:
- Phase I Dose Escalation: * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 1 AMD3100 dose = 80 mcg/kg/d
  Dose Level 2 AMD3100 dose = 160 mcg/kg/d
  Dose Level 3 AMD3100 dose = 240 mcg/kg/d
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 12
mcg/kg | 240

2. Primary Outcome: Phase II Only: Complete Response Rate of AMD3100 + MEC
Description: Responses were assessed according to the International Working Group Criteria for AML. All patients who received at least one dose of AMD3100 were considered evaluable for response.
  Response rate was the rate of complete remission plus complete remission with incomplete blood count recovery (CR + CRi).
Time Frame: 42 days
Measure: Number; unit: percentage of participants
Groups:
- Total: Phase II Dose Patients
Arm/Group | First Relapse, First Salvage | Primary Refractory | >= Second Relapse/Salvage | Total
Number analyzed (Participants) | 32 | 10 | 4 | 46
percentage of participants
  CR + CRi | 56 | 20 | 25 | 46
  CR only | 47 | 20 | 25 | 39

3. Primary Outcome: Ability of AMD3100 + MEC to Induce dsDNA Damage and Apoptosis in Leukemic Blasts From Bone Marrow or Peripheral Blood Fractions
Time Frame: 42 days
Population: This outcome was not analyzed as data was not collected.
Arm/Group | Phase I Dose Escalation/Phase II Dose Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Tolerability of AMD3100 + MEC.
Description: Treatment related mortality (deaths occurring during treatment)
Time Frame: 42 days
Population: The 46 patients include the 6 patients treated on Dose Level 3 of the Phase I portion of the study.
Measure: Number; unit: participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 46
participants
  Sepsis | 2
  Adverse transfusion reaction w/febrile neutropenia | 1

5. Secondary Outcome: Time to Neutrophil Recovery
Description: Defined as the date of the first dose of AMD3100 to the date that the absolute neutrophil count >1,000 cells/mm^3.
Time Frame: 42 days
Population: This analysis includes patients who achieved a CR or a CRi.
Measure: Median (Full Range); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 21
days | 28 [21 to 46]

6. Secondary Outcome: Time to Platelet Recovery
Description: Defined as the date of the first dose of AMD3100 to the date that the platelet count is >100,000/mm3 in the absence of platelet transfusions.
Time Frame: 42 days
Population: This analysis includes patients who achieved a CR.
Measure: Median (Full Range); unit: days
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 18
days | 28.5 [16 to 42]

7. Secondary Outcome: Characterize the Mobilization of Leukemic Cells With AMD3100 by Measuring the Peak Mobilization of Total Leukocytes (Phase I)
Description: Measured at 0 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours after AMD3100 dose on Day 0.
  Characterization of the mobilized cells as well as the kinetics of mobilization will be determined by analyzing the surface expression of mobilized cells by flow cytometry at the specified time points in conjunction with their total leukocyte count from the patient's CBC.
Time Frame: Day 0
Measure: Median (Full Range); unit: cells x 10^3/microliter
Groups:
- Phase I Dose Escalation - Dose Level 1: * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 1 AMD3100 dose = 80 mcg/kg/d
- Phase I Dose Escalation - Dose Level 2: * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 2 AMD3100 dose = 160 mcg/kg/d
- Phase I Dose Escalation - Dose Level 3: * AMD3100 SQ on days 0-5
  * Mitoxantrone on days 1-5
  * Etoposide on days 1-5
  * Cytarabine on days 1-5
  Dose Level 3 AMD3100 dose = 240 mcg/kg/d
Arm/Group | Phase I Dose Escalation - Dose Level 1 | Phase I Dose Escalation - Dose Level 2 | Phase I Dose Escalation - Dose Level 3
Number analyzed (Participants) | 3 | 3 | 6
cells x 10^3/microliter
  Total leukocytes at 0 hours | 2.5 [1.9 to 3.0] | 4.7 [2.9 to 6.1] | 3.5 [1.2 to 16.5]
  Total leukocytes at 1 hour | 4.3 [2.7 to 6.9] | 7.0 [3.9 to 10.8] | 6.4 [3.4 to 24.5]
  Total leukocytes at 2 hours | 4 [3.2 to 7.9] | 8.5 [3.7 to 11.3] | 7.5 [2.0 to 27.0]
  Total leukocytes at 4 hours | 4.7 [3.4 to 10.8] | 9.4 [3.8 to 12.1] | 8.3 [2.0 to 38.6]
  Total leukocytes at 6 hours | 4.8 [3.9 to 17.0] | 11.3 [4.3 to 14.3] | 9.5 [2.1 to 32]
  Total leukocytes at 8 hours | 4.5 [3.6 to 11.5] | 12.0 [4.4 to 16.3] | 8.9 [2.3 to 39.0]
  Total leukocytes at 12 hours | 5.1 [2.8 to 13.2] | 12.1 [5.1 to 16.0] | 7.8 [2.0 to 38.9]
  Total leukocytes at 24 hours | 4.3 [1.7 to 8.1] | 7.9 [3.4 to 11.7] | 5.8 [1.5 to 22.2]

8. Secondary Outcome: Characterize the Mobilization of Leukemic Cells With AMD3100 by Measuring the Peak Mobilization of AML Blasts (Phase I)
Description: Measured at 0 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours after AMD3100 dose on Day 0.
Time Frame: Day 0
Measure: Median (Full Range); unit: percentage of AML blasts
Arm/Group | Phase I Dose Escalation - Dose Level 1 | Phase I Dose Escalation - Dose Level 2 | Phase I Dose Escalation - Dose Level 3
Number analyzed (Participants) | 3 | 3 | 6
percentage of AML blasts
  AML blasts at 0 hours | 46.0 [2.0 to 54.0] | 4.0 [NA to NA] — The AML blasts at 0 hour was not performed on 2 out of the 3 patients. | 43.5 [10.0 to 77.0]
  AML blasts at 1 hour | 26.0 [5.0 to 34.0] | 9.0 [NA to NA] — The AML blasts at 0 hour was not performed on 2 out of the 3 patients. | 30.5 [9.0 to 68.0]
  AML blasts at 2 hours | 26.0 [3.0 to 40.0] | 37.5 [3.0 to 72.0] | 32.5 [5.0 to 67.0]
  AML blasts at 4 hours | 37.0 [4.0 to 46.0] | 16.0 [1.0 to 64.0] | 30.0 [4.0 to 60.0]
  AML blasts at 6 hours | 31.0 [2.0 to 53.0] | 14.0 [2.0 to 63.0] | 27.0 [9.0 to 74.0]
  AML blasts at 8 hours | 32.0 [5.0 to 52.0] | 19.0 [6.0 to 67.0] | 26.0 [8.0 to 70.0]
  AML blasts at 12 hours | 27.0 [2.0 to 30.0] | 45.0 [21 to 69] | 35.0 [14.0 to 82.0]
  AML blasts at 24 hours | 35.0 [3.0 to 52.0] | 23 [13 to 33] | 55 [12 to 68]

9. Secondary Outcome: Pharmacokinetics of AMD3100 on MEC
Time Frame: Day 1 - Phase 2 only
Population: This was not performed.
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to Progression
Time Frame: Every 6 months
Population: This outcome was not analyzed instead "reason for treatment failure" was analyzed as it provided better information on why the treatment did not work.
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 0

11. Secondary Outcome: Treatment Failure
Description: Treatment failures includes those patients for whom treatment has failed to achieve a CR or a CRi.
Time Frame: 42 days
Measure: Number; unit: participants
Arm/Group | First Relapse, First Salvage | Primary Refractory | >= Second Relapse/Salvage | Total
Number analyzed (Participants) | 14 | 8 | 3 | 25
participants
  Persistent leukemia | 12 | 6 | 3 | 21
  Death during aplasia | 1 | 2 | 0 | 3
  Unknown | 1 | 0 | 0 | 1

12. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 46
percentage of participants | 37

13. Secondary Outcome: Relapse-free Survival
Description: This is determined only for patients achieving a complete remission. Defined as the interval from the date of the first documentation of a leukemia free state to date of recurrence or death due to any cause.
  Kaplain-Meier estimate was used.
Time Frame: 1 year
Population: This excludes the 25 participants who had treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 21
percentage of participants | 42.9

ADVERSE EVENTS:
Time Frame: Adverse event assessment was collected from start of treatment for 42 days
Description: The adverse events are not split into Phase I Dose Escalation portion and the Phase II Dose Treatment portion instead all events are reported as a whole.
Arm/Group | Phase I Dose Escalation (Dose Level 1) | Phase I Dose Escalation (Dose Level 2) | Phase II Dose Treatment (Dose Level 3)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 3/46
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation (Dose Level 1) (N=3) | Phase I Dose Escalation (Dose Level 2) (N=3) | Phase II Dose Treatment (Dose Level 3) (N=46)
Allergic reaction - platelet transfusion (Immune system disorders) | 0 | 0 | 1 — Grade 5 - unlikely related
Hypotension (Cardiac disorders) | 0 | 0 | 1 — Unrelated
Infection-other (gram negative sepsis) (Infections and infestations) | 0 | 0 | 1 — Grade 5 unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation (Dose Level 1) (N=3) | Phase I Dose Escalation (Dose Level 2) (N=3) | Phase II Dose Treatment (Dose Level 3) (N=46)
ALT (Investigations) | 1 | 0 | 14
AST (Investigations) | 0 | 1 | 11
Abdominal cramping (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 10
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 2
Alkaline phosphatase (Investigations) | 0 | 0 | 20
Allergic reaction - NOS (Immune system disorders) | 1 | 0 | 0
Allergic reaction - general itching during transfusion (Immune system disorders) | 1 | 1 | 0
Allergic reaction - platelet transfusion (Immune system disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 25
Anxiety (Psychiatric disorders) | 2 | 3 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 8
Bilateral extremity echymosis (General disorders) | 0 | 0 | 1
Bilateral extremity petichiae (General disorders) | 0 | 0 | 2
Bladder spasms (Renal and urinary disorders) | 1 | 0 | 0
Blurred vison (Eye disorders) | 1 | 0 | 5
Bone marrow biopsy site pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2 | 8
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 2
Bumps on legs and arms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Catheter site insertion pain (Renal and urinary disorders) | 1 | 1 | 3
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 4
Chills (General disorders) | 0 | 1 | 6
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0
Coccyx pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Cognitive disturbance - lethargy (Nervous system disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis, infectious - clostridium difficile (Infections and infestations) | 0 | 0 | 4
Confusion (Psychiatric disorders) | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 2 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 13
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 4
Diaphoresis (General disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 26
Distension (Gastrointestinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 10
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 7
Edema limbs (General disorders) | 1 | 1 | 17
Edema trunk (General disorders) | 0 | 0 | 2
Epigastric pain (Gastrointestinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Esophagus pain (Gastrointestinal disorders) | 1 | 0 | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Facial pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 31
Fever (General disorders) | 0 | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized edema (General disorders) | 0 | 0 | 3
Generalized joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized pain (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 19
Heartburn (Gastrointestinal disorders) | 1 | 1 | 3
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 2
Hematoma (General disorders) | 0 | 0 | 4 — right arm and central line placement
Hemoglobin (Investigations) | 3 | 2 | 17
Hemorrhage - eye (Eye disorders) | 1 | 0 | 2
Hemorrhage - nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Hemorrhoidal pain (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Hyperbilirubinemia (Investigations) | 0 | 0 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypernatremia (Investigations) | 1 | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1 | 11
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminemia (Investigations) | 2 | 3 | 17
Hypocalcemia (Investigations) | 3 | 1 | 20
Hypokalemia (Investigations) | 2 | 1 | 11
Hyponatremia (Investigations) | 3 | 1 | 7
Hypophosphatemia (Investigations) | 2 | 1 | 6
Hypotension (Cardiac disorders) | 2 | 0 | 10
Hypothermia (General disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Incisional pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 3
Incontinence - secondary to urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Indigestion (Gastrointestinal disorders) | 1 | 0 | 0
Infection, gram positive cocci (Infections and infestations) | 0 | 0 | 1
Injection site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injection site reaction (General disorders) | 2 | 0 | 7
Insomnia (Psychiatric disorders) | 0 | 1 | 14
Itching (pruritus) (Skin and subcutaneous tissue disorders) | 2 | 0 | 10
Jaundice - right eye (Hepatobiliary disorders) | 0 | 0 | 1
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Left arm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Left elbow pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Left lower abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Leukocytes (Investigations) | 3 | 3 | 38
Lip swelling (General disorders) | 0 | 0 | 1
Liver abcess (Infections and infestations) | 0 | 0 | 1
Lower back wound pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Lymphopenia (Investigations) | 0 | 0 | 2
Mood alteration (not specified) (Psychiatric disorders) | 0 | 0 | 1
Mouth pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mouth pain - right side (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mucositis (oral and stomach) (Gastrointestinal disorders) | 1 | 2 | 33
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness - generalized (Musculoskeletal and connective tissue disorders) | 1 | 0 | 24
Nasal/paranasal reactions - sinusitis (Infections and infestations) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 33
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Neuropathy (not specified) (Nervous system disorders) | 0 | 0 | 1
Neuropathy - bilateral feet (Nervous system disorders) | 0 | 0 | 2
Neuropathy - bilateral hands (Nervous system disorders) | 0 | 0 | 1
Neuropathy - face (Nervous system disorders) | 1 | 0 | 1
Neuropathy - left eye droop (Nervous system disorders) | 0 | 0 | 1
Neuropathy - left hand (Nervous system disorders) | 0 | 0 | 1
Neuropathy - right ankle (Nervous system disorders) | 0 | 0 | 1
Neuropathy - toes (Nervous system disorders) | 0 | 0 | 3
Neutrophils (Investigations) | 3 | 1 | 21
Opportunistic infection (pneumonia NOS) (Infections and infestations) | 0 | 1 | 2
Opportunistic infection - urinary tract (Infections and infestations) | 1 | 0 | 1
Opportunistic infection, nasal (Infections and infestations) | 0 | 0 | 1
Pain upon inspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Perianal pain (Gastrointestinal disorders) | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Petichiae (General disorders) | 0 | 0 | 6
Pilonidal cyst (Injury, poisoning and procedural complications) | 0 | 0 | 1
Platelets (Investigations) | 1 | 2 | 23
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 10 — Includes undefined rash, vaginal, lower extremities, left arm, and bilateral arms.
Red and swollen left labia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Restless leg syndrome (Nervous system disorders) | 0 | 0 | 1
Rib pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right arm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right ear pain (Ear and labyrinth disorders) | 0 | 2 | 1
Right forearm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right head and neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Right side pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Right upper quadrant pain (Gastrointestinal disorders) | 0 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2 | 29
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Taste alteration (Gastrointestinal disorders) | 0 | 0 | 4
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Tooth pain (General disorders) | 0 | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 3
Urinary hesitancy (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 2
Vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Vasovagal episode (Cardiac disorders) | 0 | 1 | 0
Vision - floaters (Eye disorders) | 0 | 0 | 2
Visual changes (Eye disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 17
Weight loss (Gastrointestinal disorders) | 0 | 0 | 1
Wound - coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weakness (General disorders) | 0 | 0 | 0
Infection - gram negative sepsis (Infections and infestations) | 0 | 0 | 1
Infection - gram negative bacilli (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes